| GCS Co., Ltd. | GANA X <sup>®</sup><br>CIP #21E0805 | Final version 3.0<br>Date: 07/04/2022 | Page 1/5 |
|---|---|---|---|
|---|---|---|---|

## **SUMMARY OF THE CLINICAL INVESTIGATION PLAN # 21E0805**

| ANSM registration #: | 2021-A02728-33 |
|---|---|
| Clinical investigation plan #: | 21E0805 |
| Title of the clinical investigation: | CLINICAL STUDY FOR THE EFFECTIVENESS OF USE OF AN INJECTABLE MEDICAL DEVICE GANA X® IN THE TREATMENT OF BUTTOCKS VOLUME DEPRESSION |
| Sponsor: | GCS Co., Ltd. 1008 Ho, Sunil Technopia Bldg, 555 Dunchon-daero Jungwon-gu, Seongnam-si, Gyeonggi-do KOREA |
| Development phase | Post market study Interventional Device used according to Instruction For Use (IFU) |
| Objectives: | The primary objective is to evaluate the effectiveness of Gana X <sup>®</sup> in improving buttocks volume 6 months after treatment. |
| | <ul> <li>The secondary objectives of the study are:</li> <li>to evaluate the effectiveness of Gana X® in improving buttocks volume 1¹¹², 9, 12, 18 and 24 months after treatment.</li> <li>to evaluate the effectiveness of Gana X® on the global aesthetic improvement of buttocks 1¹¹², 6, 9, 12, 18, 24 months after treatment as rated by the evaluator.</li> <li>to evaluate the effectiveness of Gana X® on the global aesthetic improvement of buttocks 1¹¹², 6, 9 12, 18, 24 months after treatment as rated by the subjects.</li> <li>To evaluate the subject satisfaction with Gana X® 1¹¹², 6, 9, 12, 18 and 24 months after treatment.</li> <li>To evaluate the injector satisfaction with Gana X® after initial and touch-up injection if applicable.</li> <li>To evaluate the safety of Gana X®.</li> </ul> |
| Design: | The study will be: In open, Single center. |
| Planned Sample Size: | 55 subjects included. |
| Number of investigational study sites: | 1 site (France). |
| Inclusion criteria: | <ol> <li>Healthy Subject.</li> <li>Sex: male or female.</li> <li>Age: between 18 and 65 years.</li> <li>Subject with mild to moderate buttock volume depression and/or seeking buttocks volume augmentation based on investigator evaluation.</li> <li>Subject willing to abstain from other body contouring procedures during the whole study period.</li> <li>Subject psychologically able to understand the study related information and to give a written informed consent.</li> <li>Subject having given freely and expressly his/her informed consent.</li> <li>Subject willing to have photographs taken.</li> </ol> |

| GCS Co., Ltd. | GANA X <sup>®</sup><br>CIP #21E0805 | Final version 3.0<br>Date: 07/04/2022 | Page 2/5 |
|---|---|---|---|
| | 10. Female regimen | 9. Subject affiliated to a health social security system. 10. Female of childbearing potential should use a contraceptive regimen recognized as effective since at least 12 weeks before screening visit and during the whole study period. | |
| Exclusion criteria: | year or p 2. Excessiv 3. Excessiv 4. Severe b 5. Subject administi 6. Subject p who is in 8. Subject participar previous participar participar participar participar participar participar | planning a pregnancy during re subcutaneous fat in the are subcutaneous fat in the are subcutaneous fat in the are subcutaneous fat in the are subcutaneous fat in the are subcutocks ptosis. Who had been deprive rative or legal decision or win a social or sanitary estable participation to another result an exclusion period of one having already received 4 tion in research involving months or exceeding the tion in the present study. Suspected to be non-contror's judgment. Suffering from a severe or puthology that may interfere sults. With known history of or subcord in the present study of cellulitis, streeumatic fever or recurrent elematic fever with heart corn suffering from inflammus disorders in or near the excema, atopic dermatitis with an abscess, unhealed erous lesion on the studied in the prone to develop inflamment of the test of the | trea to be treated. be treated. and of their freedom by ho is under guardianship. Ishment earch on human beings or 500 euros indemnities for human beings in the 12 ese 4500 euros with his mpliant according to the progressive disease or any with the evaluation of the suffering from autoimmune reptococcal disease, such as sore throats and in case of mplications. Inatory and/or infectious studied zones (e.g. acne, ). Wound, or a cancerous or zone. Inatory skin conditions or ers. In proposed |

Buttocks implants;

| GCS Co., Ltd. | GANA X <sup>®</sup><br>CIP #21E0805 | Final version 3.0<br>Date: 07/04/2022 | Page 3/5 |
|---|---|---|---|
| | fillers Inject 1 Inject 23. Subject hother hor visit. 24. Subject inflamma antiplatel prolong because in systemic Antihologian in Immurprior Retirement and to the subjection of the subject of the | fillers or autologous fat injections); Injections for the treatment of cellulitis. 23. Subject having started or changed her oral contraceptive or any other hormonal treatment during 12 weeks prior to screening visit. 24. Subject using medication such as aspirin, nonsteroidal anti-inflammatory drugs (NSAID) (ibuprofen, naproxen,), antiplatelet agents, anticoagulants or other substances known to prolong bleeding time within 1 week prior to injection visits. 25. Subject undergoing a topical treatment on the test area or a systemic treatment: Antihistamines during the 2 weeks prior to injections visits (D0 and touch-up visit). Immunosuppressors and/or corticoids during the 4 weeks prior to injections visits (D0 and touch-up visit). Retinoids during the 6 months prior to injections visits (D0 and touch-up visit). 26. Intensive exposure to sunlight or UV-rays within the month before injection visits and one month after. 27. Subject planning to loss or gain weight for the duration of the | |
| | | study. 28. Subject planning to change her/his life habits during the study. | |
| Investigational device Name / code Classification Ingredient Galenic form Administration route | Gana X® Class III med Poly-L-Lactic Mannitol. Sterile freeze | | |
| Endpoints: | | tiveness endpoint: | |
| | treatment usi | Mean change in buttocks volume from baseline to 6 months after treatment using fringe projection system. Secondary effectiveness endpoints: | |
| | 18 a syste - GAIS treati responsimpro GAIS - GAIS treati - Prop mont - Inject and the Secondary satisfactions | and 24 months after treatment. So responder rates 11/2, 6, 9, ment as assessed by an inconder is defined as a subjectived" or "Very much important as assessed by the subjection of satisfied subjections after treatment using a control to satisfaction regarding ouch-up injection using a condense of the safety endpoints: all device safety will be | s 1 <sup>1/2</sup> , 6, 9, 12, 18 and 24 questionnaire. injection quality after initial |

| GCS Co., Ltd. | GANA X <sup>®</sup><br>CIP #21E0805 | Final version 3.0<br>Date: 07/04/2022 | Page 4/5 |
|---|---|---|---|
|---|---|---|---|

| | The state by the Secreticator Orbitator Street 10Ds and AFe Se |
|---|---|
| | the study by the investigator. Subjects will record ISRs and AEs in their subject diaries. |
| Study Procedures: | A screening visit will allow to inform and preselect the subjects. |
| | On D0, fringe projection acquisitions and photographs will be done before injection. Eligible subjects will receive a first injection of the investigational device. Immediately after injection, injector's treatment satisfaction will be collected. Investigator evaluator will collect AEs and ISRs immediately after injection. |
| | A month and a half after initial injection (M1 <sup>1/2</sup> ), GAIS scoring, fringe projection acquisitions and photographs will be done before touch-up injection (if applicable). A touch-up injection will be made if necessary, according to injector and subject opinion. Investigator evaluator will collect AEs and ISRs before and after touch-up if applicable. Subject's treatment satisfaction and injector's treatment satisfaction (if applicable) will be collected. |
| | Six (M6), nine (M9), twelve (M12), eighteen (M18) and twenty-four (M24) months after initial injection, effectiveness scoring (GAIS scale), fringe projection acquisitions and photographs will be done. Subject's treatment satisfaction will be collected. Investigator evaluator will collect AEs and ISRs |
| Statistical methods: | For the primary evaluation criterion: |
| | The primary endpoint is the mean change in buttocks volume from baseline to 6 months after treatment using fringe projection system. Descriptive statistics for quantitative data (N, mean, standard deviation, minimum and maximum) will be presented at D0 before injection and M6. |
| | Inferential analysis: |
| | A Wilcoxon signed rank test, or a paired t test will be applied to evaluate the change from baseline (D0 before injection) to M6. The normality assumption will be tested using a Shapiro Wilk test ( $\alpha$ =0.01). The bilateral approach will be used. For the secondary evaluation criteria: |
| | All the variables will be described using adapted statistics according to their type (quantitative data or qualitative data). For quantitative data a Wilcoxon or paired t test will be applied to assess the change from baseline. |
| | The bilateral approach will be used with a significance level of 0.05. |
| Foreseen study duration: | Clinical investigation beginning: Q1 2022 |
| | Clinical investigation end: Q3 2024 |
| | Inclusion duration: Maximum 6 months |
| | Clinical investigation global duration: 30 months |
| | Duration by subject: 24 months + screening period |

| GCS Co., Ltd. | GANA X <sup>®</sup><br>CIP #21E0805 | Final version 3.0<br>Date: 07/04/2022 | Page 5/5 |
|---|---|---|---|
|---|---|---|---|

## **FLOW-CHART**

| Procedure | Visit 1<br>Screening | Visit 2<br>Day 0 | Visit 3<br>M1 <sup>1/2</sup> | Visit 4<br>M6 | Visit 5<br>M9 | Visit 6<br>M12 | Visit 7<br>M18 | Visit 8<br>M24 |
|---|---|---|---|---|---|---|---|---|
| Days | D-X | D0 | D40 ± 2 | D160 ± | D270<br>±4 | D365 ± 7 | D540 ±<br>14 | D730 ± 14 |
| Informed consent form signature | • | | | | | | | |
| Medical examination | • | | | | | | | |
| Medical history and previous and concomitant treatments collection | • | | | | | | | |
| Checking of the inclusion and exclusion criteria | • | | | | | | | |
| Pregnancy test | | ●p | ●b | | | | | |
| Confirmation of eligibility | | ●p | | | | | | |
| Photographs | | <b>●</b> b | ●b | • | • | • | • | • |
| Fringe projection acquisitions (2 areas) | | <b>●</b> b | <b>●</b> b | • | • | • | • | • |
| Injection + anaesthesia (if necessary) | | • | ●Touch up | | | | | |
| GAIS live assessment by an independent evaluator | | | <b>●</b> b | • | • | • | • | • |
| GAIS assessment by the subjects | | | <b>●</b> b | • | • | • | • | • |
| Subjective evaluation questionnaire for subjects | | | <b>●</b> b | • | • | • | • | • |
| ISR live assessment by an independent evaluator | | <b>—</b> а | ●b+a | • | • | • | • | • |
| ISR assessment by the subjects | | Completed each day during 4 weeks after injection at home by the subject. | | at home | | | | |
| Subjective evaluation questionnaire for injector | | <b>•</b> а | ●a | | | | | _ |
| AE and concomitant treatments and procedures collection | • | • | • | • | • | • | • | • |
| Study end | | | | | | | | • |

Keys: b: Before injection; a: After injection